CLINICAL TRIAL: NCT05393011
Title: Vitamin D and Some Antioxidants and Trace Elements Levels in Women: Relationship With I.V.F Outcomes
Brief Title: Relationship Between Some Vitamins and Antioxidants With in Vitro Fertilization Outcomes
Status: Completed | Type: Observational
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Other Study IDs: UDFP-Biochemistry-01-2022
Record Dates: First submitted 2022-05-23; First posted 2022-05-26 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: In Vitro Fertilization; Infertility
Keywords: Vitamin D; Vitamin E; Zinc; Glutathione peroxidase
MeSH Terms: conditions — Infertility | interventions — Chorionic Gonadotropin

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

GROUPS / COHORTS (2):
- Pregnant group: A female is considered pregnant when an explicit gestational sac inside the uterus is seen by ultrasound 4 weeks after embryo transfer.
  Interventions: Drug: human chorionic gonadotropin
- Non-pregnant group: A female is considered not pregnant when no explicit gestational sac is seen inside the uterus by ultrasound 4 weeks after embryo transfer.
  Interventions: Drug: human chorionic gonadotropin

INTERVENTIONS:
Drug: human chorionic gonadotropin — 10000 IU when at least three follicles become more than 16 mm
  Other Names: Chorex

SUMMARY:
observation of females condition will getting pregnant by undergoing assisted reproductive technologies, the most important of which is the in vitro fertilization (IVF), where blood and follicular fluid samples are collected from them at the same stage of in vitro fertilization, and then monitor the IVF outcomes until pregnancy occurs or not, based on blood tests. The levels of interested markers in blood and follicular fluid samples of the study individuals are assayed in order to compare these levels with the egg criteria such as egg number and maturation rate and finally compare the results with occurrence or absence of pregnancy.

DETAILED DESCRIPTION:
Vitamin D, vitamin E, zinc and glutathione peroxidase will be measured in blood and follicular fluid samples of study subjects for women undergoing in vitro fertilization after monitoring their health for two to three months before beginning the first stage of in vitro fertilization. Once start the ovulation induction protocol, which is the first stage of in vitro fertilization, we will monitor all the results from the number of eggs and follicles, their diameter, the thickness of the endometrium, the number of mature eggs, the egg maturation rate and fertilization rate to the occurrence of biochemical pregnancy or not later, based on the blood Human chorionic gonadotropin (hCG) levels two weeks after the embryos transfer to the uterus. The patient is monitored until clinical pregnancy is complete or not. On the other hand, we will later compare the levels of studied parameters with the aforementioned egg quality criteria and with the clinical pregnancy rate of the study group in order to understand the relationship between these studied parameters and the occurrence of pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Cases of Healthy women (in terms of reproductive function).
* Aged between 20-40 years and were close in terms of education, nutrition, and social status.
* Explicit male factor such as Oligospermia, Azoospermia, Asthenozoospermia, or TESA (Testicular Sperm Aspiration), ensuring that there is no fertility-interfering female factor.
* Undergoing long Gonadotropin-releasing hormone (GnRH) agonist down-regulation protocol.

Exclusion Criteria:

* Cases classified by the specialist clinician as a female factor such as PCOs (Polycystic Ovary Syndrome), Uterine Fibroids, Uterine Infections, Uterine Adhesions, and Endometriosis.
* Compound cases.
* Sex selection cases.
* Undergoing short GnRH agonist or antagonist protocol.
* Women aged under 20 or above 40.
* Women who took nutritional supplements, for at least two to three months before the egg retrieval procedure.
* Smokers.
* Cases with the following medical conditions: Tumors, Diabetes, Multiple sclerosis, Autoimmune Diseases, Liver or Kidney Disorders, Cushing's Syndrome, and women who take chronic medications

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Females attending Orient Fertility and Genetics Hospital for infertility treatment or pregnancy assistance
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2017-08-20 (Actual); Primary Completion 2020-08-02 (Actual); Study Completion 2021-08-15 (Actual)

PRIMARY OUTCOMES:
Blood and follicular fluid vitamin D concentrations | Immediately after oocyte retrieval
  Blood and Follicular fluid samples will be obtained on the day of oocyte retrieval, then they will be centrifuged to eliminate cellular elements and debris. After that, the supernatants will be frozen at -80 until later assayed
Blood and follicular fluid vitamin E concentrations | Immediately after oocyte retrieval
  Blood and Follicular fluid samples will be obtained on the day of oocyte retrieval, then they will be centrifuged to eliminate cellular elements and debris. After that, the supernatants will be frozen at -80 until later assayed
Blood and follicular fluid zinc concentrations | Immediately after oocyte retrieval
  Blood and Follicular fluid samples will be obtained on the day of oocyte retrieval, then they will be centrifuged to eliminate cellular elements and debris. After that, the supernatants will be frozen at -80 until later assayed
Blood and follicular fluid glutathione peroxidase concentrations | Immediately after oocyte retrieval
  Blood and Follicular fluid samples will be obtained on the day of oocyte retrieval, then they will be centrifuged to eliminate cellular elements and debris. After that, the supernatants will be frozen at -80 until later assayed

SECONDARY OUTCOMES:
Number of oocytes retrieved | Immediately after oocyte retrieval
  The oocytes will be retrieved by transvaginal ultrasound-guided follicle aspiration after ovulation trigger
Number of Metaphase II Oocytes (MII) | Within two hours after oocyte retrieval
  The oocyte maturity will be assessed using Nikon SMZ1500 stereoscope
Maturation Rate% | Within two hours after oocyte retrieval
  Maturation Rate is calculated by dividing the number of mature (MII) oocytes by the number of retrieved oocytes
Fertilization Rate% | 16-18 hours after microinjection
  Fertilization Rate is calculated by dividing the number of obtained zygote (2PN) by the number of injected oocytes
Embryo Quality | Day of transfer (2 or 3 days after microinjection)
  Embryos are assessed using Nikon SMZ1500 stereoscope
Biochemical Pregnancy Rate% | 2 weeks after embryo transfer
  Biochemical pregnancy is defined as a positive serum beta-hCG pregnancy test after 2 weeks of embryo transfer. The biochemical pregnancy rate is calculated by dividing the number of women who are biochemically pregnant by the number of women who have at least 1 embryo transferred
Clinical Pregnancy Rate% (Per Embryo Transfer) | 4 weeks after embryo transfer
  weeks of embryo transfer. The clinical pregnancy rate is calculated as by dividing the number of women who are clinically pregnant divided by the number of women who have at least 1 embryo transferred

CONTACTS AND LOCATIONS:
Overall Officials: Raghad MH Faisal, MD, Principal Investigator — Damascus University
Locations (2):
- Syria (2):
  - Damascus University, Damascus
  - Orient Hospital, Damascus

IPD SHARING:
Plan to Share IPD: Undecided
The study samples will be collected from female attending Orient Hospital (assisted reproduction and genetics) in order to carry out the in vitro fertilization process after obtaining the approval of the ethical committee of Damascus University, They will be informed with their husbands of the research objectives and sign the approve consent

REFERENCES:
- [Background] Revelli A, Delle Piane L, Casano S, Molinari E, Massobrio M, Rinaudo P. Follicular fluid content and oocyte quality: from single biochemical markers to metabolomics. Reprod Biol Endocrinol. 2009 May 4;7:40. doi: 10.1186/1477-7827-7-40. PMID 19413899
- [Background] Lambalk CB, Banga FR, Huirne JA, Toftager M, Pinborg A, Homburg R, van der Veen F, van Wely M. GnRH antagonist versus long agonist protocols in IVF: a systematic review and meta-analysis accounting for patient type. Hum Reprod Update. 2017 Sep 1;23(5):560-579. doi: 10.1093/humupd/dmx017. PMID 28903472
- [Background] Aramesh S, Alifarja T, Jannesar R, Ghaffari P, Vanda R, Bazarganipour F. Does vitamin D supplementation improve ovarian reserve in women with diminished ovarian reserve and vitamin D deficiency: a before-and-after intervention study. BMC Endocr Disord. 2021 Jun 21;21(1):126. doi: 10.1186/s12902-021-00786-7. PMID 34154571
- [Background] Liu X, Zhang W, Xu Y, Chu Y, Wang X, Li Q, Ma Z, Liu Z, Wan Y. Effect of vitamin D status on normal fertilization rate following in vitro fertilization. Reprod Biol Endocrinol. 2019 Jul 18;17(1):59. doi: 10.1186/s12958-019-0500-0. PMID 31319865
- [Background] Bahadori MH, Sharami SH, Fakor F, Milani F, Pourmarzi D, Dalil-Heirati SF. Level of Vitamin E in Follicular Fluid and Serum and Oocyte Morphology and Embryo Quality in Patients Undergoing IVF Treatment. J Family Reprod Health. 2017 Jun;11(2):74-81. PMID 29282414
- [Background] Janati S, Behmanesh MA, Najafzadehvarzi H, Akhundzade Z, Poormoosavi SM. Follicular Fluid Zinc Level and Oocyte Maturity and Embryo Quality in Women with Polycystic Ovary Syndrome. Int J Fertil Steril. 2021 Jul;15(3):197-201. doi: 10.22074/IJFS.2021.135426.1006. Epub 2021 Jun 22. PMID 34155866
- [Background] Zal F, Ahmadi P, Davari M, Khademi F, Jahromi MA, Anvar Z, Jahromi BN. Glutathione-dependent enzymes in the follicular fluid of the first-retrieved oocyte and their impact on oocyte and embryos in polycystic ovary syndrome: A cross-sectional study. Int J Reprod Biomed. 2020 Jun 30;18(6):415-424. doi: 10.18502/ijrm.v13i6.7283. eCollection 2020 Jun. PMID 32754677